CLINICAL TRIAL: NCT02764619
Title: Phase 3, Prospective, Randomized, Double-blinded, Placebo-controlled Study to Evaluate Efficacy of add-on Therapy With Spironolactone to Reduce Diffuse Myocardial Fibrosis Thus Preventing Recurrent Episodes of Atrial Fibrillation in Patients With Paroxysmal or Persistent Atrial Fibrillation and Preserved Ejection Fraction Compared to Usual Care.
Brief Title: Inhibition of Aldosterone to Reduce Myocardial Diffuse Fibrosis in Patients With Paroxysmal and Persistent Atrial Fibrillation in Preventing Recurrent Episodes of Atrial Fibrillation
Acronym: INSPIRE-AF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Svendborg Hospital (Other)
Collaborators: Region of Southern Denmark (Other); Takeda (Industry)
Responsible Party: Principal Investigator, Dragana Rujic, MD, ph.d.-student, Svendborg Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPI-IIT-001
Record Dates: First submitted 2016-03-27; First posted 2016-05-06 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Atrial Fibrillation
Keywords: Upstream therapy, spironolactone; Atrial remodelling; Modified look-locker inversion recover (MOLLI) sequences; T1 mapping; Diffuse myocardial fibrosis
MeSH Terms: conditions — Atrial Fibrillation | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aldo group (Active Comparator): Fixed dose of spironolactone, Spirix (Takeda Pharma A/S), 25 mg once daily, added to optimal medical treatment (usual care) for atrial fibrillation.
  Interventions: Drug: Spironolactone
- Control group (Placebo Comparator): Matched placebo, 1 pill once daily, added to optimal medical treatment (usual care) for atrial fibrillation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone
  Other Names: Spirix; Spiron; Hexalacton
  Arms: Aldo group
Drug: Placebo
  Arms: Control group

SUMMARY:
A randomized, double-blinded, placebo-controlled study to evaluate the effect of spironolactone in addition to conventional treatment compared with placebo in patients with paroxysmal and persistent atrial fibrillation with preserved left ventricular ejection fraction by T1 mapping, structure and function of left atrium and ventricle assessed by transthoracic echocardiography and cardiac magnetic resonance (CMR), the number of recurrent episodes of atrial fibrillation and biomarkers measured in blood.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common sustained cardiac arrhythmia present in 1% of population under 60 years of age and reaching up to 15 % at 80 years. Due to demographic changes in the Danish population, the incidence and prevalence of AF is expected to double within the next 30 years. Furthermore a number of diseases which are associated with a higher prevalence of AF such as ischemic heart disease, valvular heart disease, diabetes mellitus and hypertension are also expected to increase in prevalence due to the aging population which will contribute to an increased incidence of AF. AF increases mortality and causes important morbidity, mainly due to thromboembolic complications and increases health economic costs. Additionally, AF is associated with reduced quality of life.

The onset and maintenance of AF is highly complex and the most frequent pathoanatomic changes in AF are atrial fibrosis. In recent years, experimental and clinical studies have demonstrated that atrial remodelling and dilation in AF depending on cellular hypertrophy, fibroblast proliferation and tissue fibrosis. Atrial fibrosis leads to disruption of the electrical side-to-side junctions between muscle bundles and has potentially arrhythmogenic mechanisms. The association of atrial fibrosis and AF has been the subject of intense recent investigation, and it is now widely accepted that interstitial fibrosis creates a substrate for arrhythmia. It is believed that when atrial myocardial fibre bundles are separated by connective tissue, the conduction properties are altered because of the effects on axial resistance, leading to arrhythmia. Myocardial fibrosis is preceded by a growing activity of extracellular matrix (ECM), pro-inflammatory cytokines and at the same time more pronounced collagen (type I and III) expression. Histological studies in patients with both AF and sick sinus syndrome have shown extensive fibrosis of the atrial muscle in the sinus node and internodal tracts. These results suggest that myocardial interstitial fibrosis plays a crucial role in AF .

Recent research suggests that many of the structural and electrophysiological changes that lead to AF can be attenuated or reversed through treatment with Upstream Therapy targeting the rennin-angiotensin II-aldosterone system (RAAS). Upstream therapy such as angiotensin-converting enzyme inhibitors (ACEIs), angiotensin II receptor blockers (ARBs) and spironolactone possess antifibrotic properties, in addition, to their more well-known mechanisms of action. Most clinical trial data suggest RAAS inhibition with ACEI or ARB are associated with a lower risk of incident AF in patients with heart failure, but data from hypertension trials have been inconsistent.

Increased activation of RAAS may have a key role in the development and maintenance in AF. Especially angiotensin II and aldosterone draw attention. Aldosterone has hypertensive action, induces hypertrophy and fibrosis of cardiomyocytes and endothelium, modulating ion currents and refractoriness in the heart cycle. Arrhythmogenic aldosterone mechanisms include inhibition of noradrenalin reuptake, attenuation of baroreceptor activity, increase their sensitivity to catecholamines and reduce sinus rhythm variability. The expression of both the aldosterone receptor and angiotensin II receptors (AT1 and AT2) is increased in the atria of AF patients. For example, Boldt et al. reported a 100 % increase in AT1 receptor density in the left atrium in patients with chronic and paroxysmal AF compared to sinus rhythm . This reflects increased tissue activation of angiotensin II in fibrillating atria. Moreover, multiple studies have demonstrated a vicious cycle of RAAS in which aldosterone enhances the effects of angiotensin II, in part via an increased transcription of the AT1 receptor, whereas angiotensin II increases systemic and tissue levels of aldosterone. These findings are consistent with findings of elevated plasma levels of both angiotensin II and aldosterone during AF in a study by Goette et al. By blocking mineralocorticoid receptors with MRAs, RAAS over-activation can be diminished. Available data suggest that there are direct effects of spironolactone on the structural and electrical properties of the atria, preventing occurrence and maintenance of AF through its antifibrotic properties, as well as the indirect influence of improved control of heart failure and hypertension, both of which are known risk factors for AF.

Dabrowski et al. documented a significant reduction (p<0.0001) in the recurrence of symptomatic AF episodes in patients with symptomatic paroxysmal AF treated with spironolactone 25 mg/day compared to patients treated with enalapril or a beta-blocker. In addition, the effect of spironolactone was more prominent than that of enalapril already after 9-12 months treatment, where the effect of enalapril was less pronounced. Moreover, the addition of enalapril to spironolactone did not influence the frequency of AF recurrences.

New research acknowledges that long-term treatment with ACEI or ARB does not reliably suppress RAAS over the long term, a well-documented phenomenon known as aldosterone escape. Aldosterone is a potentially important component of RAAS, which has not been well investigated in the context of AF prevention in patients without heart failure. After a period of initial suppression, aldosterone concentrations increase to normal or above normal levels. Spironolactone can prevent aldosterone escape and prohibit fibrosis more effectively than ACEI and ARB. It was shown to reduce mortality in patients with heart failure, but data on the effect on the incidence of atrial fibrillation are still limited.

Hypothesis:

Spironolactone added to optimal medical treatment will reduce diffuse myocardial fibrosis, diminish atrial remodeling and improve function of left atrium and ventricle, thus preventing recurrent episodes of AF and decrease inflammatory biomarkers as compared with conventional treatment.

Study design: This is a prospective, randomized, double-blinded, placebo-controlled, parallel group, single center, investigator-initiated study.

The intervention group: spironolactone at a fixed dose of 25 mg per day. The control group: placebo. Patients in both groups will be treated with the study medicine throughout 12 months and additionally follow the same therapeutic recommendations according to the Danish Society of Cardiology guidelines on treatment of AF.

Comprehensive transthoracic echocardiography, 12-lead ECG, biomarkers and Holter monitoring will be performed at the time of randomization and at 6 and 12 months, respectively. Blood samples and ECG will be collected one week after the onset of treatment, and subsequently at 1, 2,3,6,9 and 12 months. During this period of 12 months, all patients will be followed for recurrence of symptomatic AF. Any relapse of symptomatic arrhythmia should be documented, if possible by 12-lead ECG or Holter monitoring. Only documented AF-recurrence by 12-lead ECG or Holter monitoring will be taken into account. CMR exams will be preformed at baseline and at 12 months, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age, male or female.
* Paroxysmal or persistent atrial fibrillation on one occasion, detected on 12-lead ECG or Holter monitoring with atrial fibrillation episode lasting ≥ 30 seconds within last 12 months prior to the screening visit.
* Women with childbearing potency must use effective contraception (e.g. implants, hormonal depot injections, combined oral contraceptives, intra-uterine devices or vasectomized partner). Men enrolled in this study must agree to use adequate barrier birth control measures during the treatment period of the study. Reliable contraception should be maintained throughout the study and for 30 days after study drug discontinuation.
* Written informed consent signed before any study-specific procedure.

Exclusion Criteria:

* Permanent AF.
* Previous radiofrequency ablation and / or previous surgical therapy of AF.
* Heart failure (New York Heart Association [NYHA] ≥ II or/and left ventricular ejection fraction [LVEF] less than 40%).
* Severe coronary artery disease (acute coronary syndrome (ACS) within 6 months prior to the screening visit, previous coronary artery bypass graft [CABG] or stabile angina pectoris classified with Canadian Cardiovascular Society [CCS] ≥II). The definition of ACS is from the current European Society of Cardiology (ESC) and American College of Cardiology (ACC) / American Heart Association (AHA) guidelines.
* Stroke or transient ischemic cerebral attack within 6 months prior to the screening visit.
* Pregnant women, breastfeeding women or women of childbearing potential not on adequate birth control.
* Presence of severe and hemodynamically significant valvular heart disease.
* Hepatic insufficiency classified as Child-Pugh B or C .
* Any disease that limits life expectancy to less than 1 year.
* Participation in another clinical trial, either within the last 30 days or ongoing.
* Morbus Addison.
* Ongoing therapy with class IC agents (flecainide, propafenone) or amiodarone, dronedarone sotalol.
* Chronic kidney disease (estimated glomerular filtration rate [eGFR] ≤ 45 ml/min/1,73 m2 [MDRD]).
* Intolerance or contradictions to spironolactone, i.e. latest product resume on Spirix®.
* Patients who are noncompliant with treatment.
* Mental disorders suspected to interact with study outcome or any other patient characteristics that may interfere with adherence to the study protocol, such as dementia, substance abuse.
* Any surgical or medical condition that in the opinion of the investigator would jeopardize the evaluation of efficacy or safety.
* Baseline serum potassium ≥ 5,0 mmol/l or serum sodium < 135 mmol/l. Note: one re-assessment of electrolytes is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2013-12; Primary Completion 2017-02 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Determine change (∆) in diffuse myocardial fibrosis between groups, assessed by cardiovascular magnetic resonance (CMR) T1 mapping. | Change from baseline at 12 months
  The study aims to non-invasively quantify extracellular volume fraction (ECV) in left atrium and ventricle as surrogate marker of diffuse myocardial fibrosis. T1 relaxation times (T1 values) will be obtained from T1 mapping. T1 values are given in [ms]. Extracellular volume fraction (ECV) will be calculated using pre-contrast and post-contrast T1 values for myocardium and blood pool (using hematocrit) using following formula: ECV = (√T1 "myocardium post-contrast" - 1 / T1 "myocardium pre-contrast") (1 / T1 "blood post-contrast" - 1 / T1 "blood pre-contrast") x (1- hematocrit). ECV is given in percentage.
Determine difference (α) in myocardial stiffness between groups, assessed by strain analysis. | At time of randomization, 6 and 12 months
  The study aims to characterize longitudinal changes in imaging characteristics.Strain is a dimensionless quantity and is produced by application of stress. It represents the fractional or percentage change from the original or unstressed dimension and includes both lengthening, or expansion (positive strains) and shortening, or compression (negative strains). Strain rate is the temporal derivative of strain and is a measure of the rate of deformation, with units of [1/s]. The strain rate is also equivalent to the shortening velocity per fiber length.
Determine difference (β) in left atrial phasic function between groups, assessed by transthoracic echocardiography. | At time of randomization and 12 months
  Left atrial phasic function is measured by the volumetric method, where LA volumes are measured at different time points of the cardiac cycle. Left atrial volumes on time curves are indexed to body surface area and are given in [mL/m2]. Speckle tracking is a technique that is complementing phasic function measures with myocardial deformation. Quantitative curves are representing all segments showing wall deformation during the cardiac cycle.

SECONDARY OUTCOMES:
Arrhythmic composite endpoint. | 12 months from randomization
  Burden of atrial fibrillation, where recurrent episodes of atrial fibrillation are documented with 12-lead ECG recordings and serial Holter monitoring. AF burden assessed as cumulative AF burden, registered on 12-lead ECG recordings and serial 48-hour Holter monitoring, where a recurrent episode of AF is defined as AF ≥ 30 seconds of duration. AF burden will also include the total duration of AF, recorded on Holter monitoring.
Life quality, assessed by SF-12. | At time of randomization and 12 months
Determine level of collagen turnover between groups, measured in blood. | At time of randomization, 6 and 12 months
  The aims of the study are:
  * To investigate whether or not the burden of diffuse myocardial fibrosis (T1 mapping) is associated with biomarkers measured in blood.
  * To investigate whether or not left atrial volume and function is associated with biomarkers measured in blood.
  Additional biomarkers may be included as the research in those fields progresses during the conduct of this clinical trial.
Adverse events | 15 months from randomization
  Adverse events (AE's) and serious adverse events (SAE's) of special interest that is hyperkalemia (serum potassium ≥ 5,5 mmol/l and serum potassium ≥ 6 mmol/l), worsening renal function (WRF) defined as a 30 % reduction in estimated glomerular filtration rate (eGFR) from baseline and gynecomastia ( Common Terminology Criteria for Adverse Events version 5.0, grade ≥ 1).

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Egstrup, Professor, Study Director — Department of Cardiovascular Research, Medical Department, Odense University Hospital, Svendborg; Dragana Rujic, MD, Ph.D.sc., Principal Investigator — Department of Cardiovascular Research, Medical Department, Odense University Hospital, Svendborg
Locations (1):
- Department of Cardiovascular Research, Medical Department, Odense University Hospital, Svendborg, Svendborg, Region Syddanmark, Denmark